CLINICAL TRIAL: NCT06846229
Title: A Cohort Study to Evaluate an Artificial Intelligence Model for Assisting Medical Decision-Making Using Real-Time Hospital-Wide Electronic Health Record Data
Brief Title: AI-Assisted Medical Decision-Making
Status: Recruiting | Type: Observational
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kang Zhang, Chief Scientist, Wenzhou Medical University
Other Study IDs: AI Prediction
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Real-world Study
Keywords: diagnosis; prediction; AI; outcome
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospital-Wide Patient Cohort
  Interventions: Other: AI-associated strategy

INTERVENTIONS:
Other: AI-associated strategy — The intervention in this study involves an AI system that leverages multimodal data fusion to support the clinical decision-making and evaluation of diseases. Patients in this cohort will undergo standard examinations, with clinical decisions guided by the recommendations generated by the AI system.

SUMMARY:
The study builds and applies an AI model to help doctors predict patient diagnoses and outcomes, such as survival or hospital stay. Real-time, multimodal data (labs, vital signs, history, imaging) from hospital records will be used. Patients will be tracked to compare the AI's performance with standard care. The goal is to improve diagnosis and treatment accuracy in a real-world, prospective study.

DETAILED DESCRIPTION:
This study aims to build and apply an artificial intelligence (AI) model to assist doctors in predicting patient diagnoses and outcomes, such as survival or hospital stay length. Patients will be enrolled across the hospital, and real-time, multimodal health data-including lab results, vital signs, medical history, and imaging-from electronic health records will be used. The study will follow participants to evaluate the AI model's performance against standard practice. The goal is to improve the accuracy and speed of diagnoses and treatments, enhancing patient care. This prospective study tests the model in real-world hospital settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to any department of the hospital (e.g., ICU, general wards, emergency, outpatient services) during the study period.
2. Patients with available real-time electronic health record (EHR) data, including at least two of the following: laboratory results, vital signs, medical history, and imaging data.

Exclusion Criteria:

Patients currently enrolled in another clinical trial that could interfere with data collection or outcomes of this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes all patients admitted to any hospital department, with real-time electronic health record data (e.g., labs, vital signs, history, imaging). Participants must consent to data collection.
Sampling Method: Non-Probability Sample
Enrollment: 50000000 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | 1 year
  AUC of the ROC curve, used to quantify diagnostic accuracy. No unit (a ratio or percentage, typically expressed as a number between 0 and 1).
Overall Hospital Resource Utilization Improvement | 1 year
  The percentage reduction in overall hospital resource use (e.g., bed days, ICU admissions, diagnostic tests) attributed to AI-assisted decision-making, expressed as a percentage.
Population-Level Diagnostic Accuracy Enhancement | 1 year
  The overall improvement in diagnostic accuracy across all hospital patients (e.g., percentage of correct diagnoses or reduction in misdiagnoses) facilitated by the AI model, expressed as a percentage or ratio.
System-Wide Reduction in Adverse Event Rates | 1 year
  The percentage reduction in major adverse events (e.g., mortality, severe complications, or prolonged stays) across all hospital patients due to AI-assisted decision-making, expressed as a percentage.

SECONDARY OUTCOMES:
Overall Improvement in Hospital Patient Outcomes | 1 year
  The aggregate improvement in key patient outcomes (e.g., mortality, morbidity, recovery rates) across the entire hospital population due to AI-assisted decision-making, expressed as a composite score or percentage.
Enhancement of Healthcare System Efficiency | 1 year
  he overall improvement in hospital operational efficiency (e.g., reduced wait times, optimized resource allocation, decreased staff workload) attributed to the AI model, expressed as a percentage or qualitative rating.
Population Health Impact Score | 1 year
  A composite score reflecting the AI model's effect on population health within the hospital's catchment area (e.g., reduced disease burden, improved chronic disease management), expressed as a standardized index or percentage change.
Long-Term Public Health Benefit Index | 1 year
  A composite index measuring the AI model's long-term contribution to public health (e.g., reduced disease prevalence, improved life expectancy), expressed as a standardized score or percentage improvement.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No